

# Global Medical Affairs

# RAD001 (Everolimus) Afinitor

Oncology Clinical Protocol CRAD001C2X01B / NCT01789281

An open-label, multi-center everolimus roll-over protocol for patients who have completed a previous Novartis-sponsored everolimus study and are judged by the investigator to benefit from continued everolimus treatment

**Authors** 

Document type Amended Protocol Version

EUDRACT number 2012-004707-12

Version number 01 (Amendment) (Clean)

Development phase IV

Document status Final

Release date 18-Mar-2016

Property of Novartis

Confidential

May not be used, divulged, published or otherwise disclosed without the consent of Novartis

Template version 19-Nov-2015

List of abbreviations 6
Glossary of terms 7
Amendment 01 (18-Mar-2016) 9
Protocol summary: 11

Background 13

Rationale 16

Study rationale and purpose 16

Rationale for dose and regimen selection \_\_\_\_\_\_\_16

Risks & Benefits 17

Definition of end of study......21

Early study termination 21

Patient population ......21

Inclusion criteria 21
Exclusion criteria 22

Ancillary treatments 24

Rescue medication 24

Objectives and endpoints 18

Treatment 23

Overview of everolimus 13

1

2

4

1.1

1.2

2.1

2.2

2.3

24

2.5

2.6

4 1

4.2

4.3

4.4

5.1

5.2

53

6.1

6.1.1

6.1.2

6.1.3

6.1.4

6.1.5

Treatment duration.

# Table of contents Table of contents List of figures List of tables 5

| | 6.2 | Dose es | scalation guidelines | 24 |
|---|---|---|---|---|
| 6.3 Dose modifications | | nodifications | 24 | |
| | | 6.3.1 | Dose modification and dose delay | 24 |
| | | 6.3.2 | Follow-up for toxicities | 25 |
| | | 6.3.3 | Anticipated risks and safety concerns of the study drug | |
| | 6.4 | Concor | nitant medications | |
| | | 6.4.1 | Permitted concomitant therapy | 26 |
| | | 6.4.2 | Permitted concomitant therapy requiring caution and/or action | |
| | | 6.4.3 | Prohibited concomitant therapy | 28 |
| | | 6.4.4 | Use of Bisphosphonates (or other concomitant agents) | |
| | 6.5 | Patient | numbering, treatment assignment or randomization | |
| | | 6.5.1 | Patient numbering | |
| | | 6.5.2 | Treatment assignment or randomization | |
| | | 6.5.3 | Treatment blinding | |
| | 6.6 | Study d | Irug preparation and dispensation | |
| | | 6.6.1 | Study treatment packaging and labeling | |
| | | 6.6.2 | Drug supply and storage | |
| | | 6.6.3 | Study drug compliance and accountability | |
| | | 6.6.4 | Disposal and destruction | 31 |
| 7 | Visit | schedule | and assessments | 31 |
| | 7.1 Study flow and visit schedule | | 31 | |
| | | 7.1.1 | Molecular pre-screening | 33 |
| | | 7.1.2 | Screening | 33 |
| | | 6.3.1 Dose modification and dose delay 6.3.2 Follow-up for toxicities 6.3.3 Anticipated risks and safety concern Concomitant medications 6.4.1 Permitted concomitant therapy 6.4.2 Permitted concomitant therapy requ 6.4.3 Prohibited concomitant therapy 6.4.4 Use of Bisphosphonates (or other concomitant numbering, treatment assignment or rat 6.5.1 Patient numbering 6.5.2 Treatment assignment or randomizat 6.5.3 Treatment blinding 6.6.1 Study drug preparation and dispensation 6.6.1 Study treatment packaging and label 6.6.2 Drug supply and storage 6.6.3 Study drug compliance and accountated 6.6.4 Disposal and destruction 6.6.5 Study flow and visit schedule 7.1.1 Molecular pre-screening 7.1.2 Screening 7.1.3 Run-in period 7.1.4 Treatment period 7.1.5 Discontinuation of study treatment 7.1.6 Follow up for safety evaluations 7.1.7 Lost to follow-up 7.1.8 Assessment types 7.2.1 Efficacy assessments 7.2.2 Safety and tolerability assessments 7.2.3 Pharmacokinetics 7.2.4 Biomarkers 7.2.5 Resource utilization 7.2.6 Patient reported outcomes | Run-in period | 33 |
| | | 7.1.4 | Treatment period | 33 |
| | | 7.1.5 | Discontinuation of study treatment | 33 |
| | | 7.1.6 | Follow up for safety evaluations | |
| | | 7.1.7 | Lost to follow-up | 35 |
| | 7.2 Assessment types | | | |
| | | | Efficacy assessments | |
| | | 7.2.2 | Safety and tolerability assessments | |
| | | 7.2.3 | Pharmacokinetics | 35 |
| | | 7.2.4 | Biomarkers | 35 |
| | | 7.2.5 | Resource utilization | |
| | | 7.2.6 | Patient reported outcomes | |
| 8 | Safet | | ring and reporting | |
| | - | | = | |

Page 4

Sample size calculation......44

10.8

| | 10.9 | Power fo | or analysis of key secondary variables | 44 |
|---|---|---|---|---|
| 11 | Ethica | ıl consider | rations and administrative procedures | 45 |
| | 11.1 | Regulato | ory and ethical compliance | 45 |
| | 11.2 | Respons | ibilities of the investigator and IRB/IEC/REB | 45 |
| | 11.3 | Informed | d consent procedures | 45 |
| | 11.4 | Disconti | nuation of the study | 46 |
| | 11.5 | Publicati | on of study protocol and results | 46 |
| | 11.6 | Study do | cumentation, record keeping and retention of documents | 46 |
| | 11.7 | Confider | ntiality of study documents and patient records | 47 |
| | 11.8 | Audits a | nd inspections | 47 |
| | 11.9 | Financia | l disclosures | 47 |
| 12 | Protoc | ol adhere | nce | 47 |
| | 12.1 | Amendn | nents to the protocol | 47 |
| 13 | Refere | | ilable upon request) | |
| | gure 4-1 | gures | Study design | 20 |
| | st of ta | ables | Objectives and related endpoints | 10 |
| | ole 6-1 | | Dose and treatment schedule | |
| | ole 6-2 | | Combination therapy dose and treatment schedule | |
| | ole 6-3 | | Clinically relevant drug interactions: inducers, and inhibitors of isoenzyme CYP3A | |
| Tal | ole 6-4 | | Clinically relevant drug interactions: substrates, inducers, inhibitors of PgP and PgP/CYP3A dual inhibitors | |
| Table 6-5 | | | Preparation and dispensing | 29 |
| Tal | ole 6-6 | | Packaging and labeling | 29 |
| Tal | ole 6-7 | | Supply and storage of study treatments | 30 |
| Table 7-1 | | | Visit evaluation schedule | 32 |

### List of abbreviations

AE Adverse Event

BSC Best Supportive Care

CRF Case Report/Record Form; the term CRF can be applied to either EDC or Paper

CRO Contract Research Organization

CSR Clinical study report
EC European Commission
IB Investigator's Brochure

ICH International Conference on Harmonization

IEC Independent Ethics Committee
IIT Investigator-initiated Trial
IRB Institutional Review Board

mTOR mammalian Target of Rapamycin

OGD&GMA Oncology Global Development and Global Medical Affairs

o.d. omnia die/once a day
PI Principal Investigator
p.o. per os/by mouth/orally
REB Research Ethics Board
SAE Serious Adverse Event

SOP Standard Operating Procedure

# **Glossary of terms**

| Assessment | A procedure used to generate data required by the study |
|---|---|
| Control drug | A study treatment used as a comparator to reduce assessment bias, preserve blinding of investigational drug, assess internal study validity, and/or evaluate comparative effects of the investigational drug |
| Cycles | Number and timing or recommended repetitions of therapy are usually expressed as number of days (e.g.: q28 days) |
| Dose level | The dose of drug given to the patient (total daily or weekly etc.) |
| Enrollment | Point/time of patient entry into the study; the point at which informed consent must be obtained (i.e. prior to starting any of the procedures described in the protocol) |
| Investigational treatment | Drug whose properties are being tested in the study as well as their associated placebo and active treatment controls (when applicable). This also includes approved drugs used outside of their indication/approved dosage, or that are tested in a fixed combination. Investigational treatment generally does not include other study treatments administered as concomitant background therapy required or allowed by the protocol when used in within approved indication/dosage |
| Medication number | A unique identifier on the label of each study treatment package which is linked to one of the treatment groups of a study |
| Other study treatment | Any drug administered to the patient as part of the required study procedures that was not included in the investigational treatment |
| Patient Number (Patient No) | A unique identifying number assigned to each patient/subject/healthy volunteer who enrolls in the study |
| Roll-over study | A roll-over study allows patients from multiple parent studies spanning multiple indications to continue to be treated within one study after the completion of the parent study(ies) |
| Stage in cancer | The extent of a cancer in the body. Staging is usually based on the size of the tumor, whether lymph nodes contain cancer, and whether the cancer has spread from the original site to other parts of the body |
| Stop study participation | Point/time at which the patient came in for a final evaluation visit or when study treatment was discontinued whichever is later |
| Study treatment | Includes any drug or combination of drugs in any study arm administered to the patient (subject) as part of the required study procedures, including placebo and active drug run-ins. |
| | In specific examples, it is important to judge investigational treatment component relationship relative to a study treatment combination; study treatment in this case refers to the investigational and non-investigational treatments in combination. |
| Study treatment discontinuation | Point/time when patient permanently stops taking study treatment for any reason |
| Supportive treatment | Refers to any treatment required by the exposure to a study treatment, e.g. premedication of vitamin supplementation and corticosteroid for pemetrexed disodium. |
| Treatment group | A treatment group defines the dose and regimen or the combination, and may consist of 1 or more cohorts. Cohorts are not expanded, new cohorts are enrolled. |

| Variable | Identifier used in the data analysis; derived directly or indirectly from data collected using specified assessments at specified timepoints |
|---|---|
| Withdrawal of consent | Withdrawal of consent occurs only when a patient does not want to participate in the study any longer, and does not want any further visits or assessments, and does not want any further study related contact |

# **Amendment 01 (18-Mar-2016)**

### **Amendment rationale**

The main purpose of the amendment is to change the primary endpoint to safety to better characterize the long-term safety of the compound. In addition, the protocol has been amended to include the collection of all AEs (including non-serious AEs) and an investigator attestation of continued clinical benefit

This roll-over study has been opened since 13-May-2013 with 32 patients enrolled and 21 patients ongoing.

# Changes to the protocol

Changes to specific sections of the protocol are shown in the track changes version of the protocol using strike through red font for deletions and red underlined for insertions.

The following changes have been implemented:

- Section 1.1: Removed the purpose of the study as this was redundant to Section 2.1.
- Section 1.2.1: Overview language updated based on IB update.
- Section 1.2.1.2: Clinical experience language updated based on IB update.
- Section 2.1: Updated purpose to reflect new primary endpoint.
- Section 2.2: Updated rationale to reflect new primary endpoint.
- Table 3-1: Updated with revised study objectives. The primary objective is to evaluate long term safety data. The secondary objective is to evaluate clinical benefit as assessed by the investigator.
- Section 4.1: Updated description of study to reflect new primary endpoint and to clarify that all adverse events and serious adverse events will be collected continuously throughout the study. Visit frequency updated to quarterly. Updated to specify that at every visit, the investigator is required to confirm that the patient continues to have clinical benefit and may continue receiving study treatment.
- Section 4.2: Updated to reflect that interim analyses are not applicable.
- Section 4.3: Updated definition of the end of study.
- Section 5.3: Updated contraception languagebased on new guidelines on pregnancy prevention.
- Section 6.1: Removed reference to drug shipments to sites.
- Section 6.1.5: Updated to specify that at every visit, the investigator is required to confirm that the patient continues to have clinical benefit and may continue receiving study treatment.
- Section 6.3.1: Added reference to IB for dose modifications.
- Section 6.3.2: Added that patients will be followed for adverse events in addition to serious adverse events.

- Section 6.3.2.1: New section added for drug-induced liver toxicity language.
- Section 6.4: Added reference to IB for use concomitant medications.
- Table 6-3: Updated inducers, and inhibitors of isoenzyme CYP3A based on IB update.
- Table 6-4: Updated substrates, inducers, inhibitors of PgP and PgP/CYP3A dual inhibitors based on IB update.
- Section 6.4.2: Updated vaccination languagebased on IB update.
- Table 6-5: Updated to reflect change to quarterly visits.
- Table 7-1: Updated to include investigator attestation of clinical benefit at every quarterly visit, collection of all adverse events, relevant medical history, monthly at home pregnancy testing for female patients of child bearing potential and the study evaluation completion eCRF page at the end of the 30 day safety follow up.
- Section 7.1.2.3: Updated to reflect collection of demographics and relevant medical history.
- Section 7.1.4: Updated to specify amount of drug supply to be provided, visits are quarterly, and that the investigator is required to confirm that the patient continues to have clinical benefit at every visit and may continue receiving study treatment.
- Section 7.1.5: Section name updated.
- Section 7.1.5.1: Section name updated in addition to adding new language.
- Section 7.1.6: Section name updated. Added stipulation that adverse events be collected.
- Section 7.1.6.1: Added new section for study evaluation completion.
- Section 7.1.7: Added Lost to follow up language.
- Section 7.2.1: Updated to specify that the investigator is required to confirm that the patient continues to have clinical benefit at every visit and may continue receiving study treatment.
- Section 7.2.2: Updated pregnancy testing language.
- Section 8: Updated with new AE/SAE reporting process.
- Section 10: Updated statistical analysis section based on revised study objectives.
- Section 11.4: Added reference to Section 4.4.
- Section 13: Removed references no longer used.

References to the parent protocol have been removed in favor of a newer source that can be used (for example, the IB), as applicable. The protocol summary has also been updated to reflect the above changes, as applicable.

A copy of this amended protocol will be sent to the Institutional Review Board (IRBs)/Independent Ethics Committee (IECs) and Health Authorities.

The changes described in this amended protocol require IRB/IEC approval prior to implementation.

# **Protocol summary:**

| Protocol summary: | |
|---|---|
| Title | An open label, multi-center everolimus roll-over protocol for patients who have completed a previous Novartis-sponsored everolimus study and are judged by the investigator to benefit from continued everolimus treatment. |
| Sponsor and Clinical Phase | Novartis, IV. |
| Investigation type | Drug. |
| Study type | Interventional. |
| Purpose and rationale | The purpose of this study is to better characterize the long- term safety of everolimus in patients who are on everolimus treatment in a Novartis-sponsored, Oncology Global Development & Global Medical Affairs (OGD&GMA) study and are benefiting from the treatment as judged by the investigator. |
| Primary Objective | To evaluate long term safety data. |
| Secondary Objectives | To evaluate clinical benefit as assessed by the investigator |
| Study design | This is a multi-center, open label study to better characterize the long-term safety of everolimus in patients being treated in current Novartis-sponsored OGD&GMA studies and who are benefiting from treatment with everolimus as judged by the investigator. There will be no screening period for this study. Eligible patients are to be consented and can start their treatment with everolimus as soon as they enter the study. All patients must report to the study site for their first visit at which time, a quarterly supply of everolimus can be dispensed to the patient/or as per local practice. Patients must return to the study center on a quarterly basis 12 weeks +/- 1 week) for resupply of study medication at which time drug dispensing information and adverse events will be collected. The patient may return to the clinic at any given time as per standard of care, however, only four study visits per year will be recorded. All adverse events and serious adverse events will be collected continuously throughout the study. Patients will continue to be treated until they are no longer benefiting from everolimus as judged by the investigator (disease progression), develop unacceptable toxicities, withdraw consent, are non-compliant to the protocol, or the patient dies, whichever comes first. A patient will reach the end of study when everolimus treatment is permanently discontinued and the end of treatment visit has been performed. All patients must be followed for adverse events and serious adverse events for 30 days after the last dose of study treatment. Following this there are no further follow-up study visits. The study is expected to remain open for 10 years or until such time that enrolled patients no longer need treatment with everolimus or are able to obtain commercial supply according to local regulations for their medical conditions. |
| Population | Male and female patients, who are currently enrolled in a Novartis-sponsored, OGD&GMA everolimus study, are benefiting from treatment with everolimus and have fulfilled all their requirements in the parent study. All objectives of the parent study must have been reached, and the study must be in the process of being completed & reported. Approximately 50 patients may enroll into this study. |
| Inclusion criteria | Patient is currently enrolled in a Novartis- sponsored, Oncology Clinical Development & Medical Affairs study receiving everolimus and has fulfilled all their requirements in the parent study. Patient is currently benefiting from the treatment with everolimus, as determined by the parent study criteria. Patient has demonstrated compliance, as assessed by the investigator, with the parent study protocol requirements. |

| Exclusion criteria | Patient has been permanently discontinued from everolimus study treatment in the parent study due any reason. |
|---|---|
| | Patient has participated in a Novartis sponsored combination trial where everolimus was dispensed in combination with unapproved or experimental treatments and is still receiving the unapproved or experimental treatment. |
| Investigational and reference therapy | Everolimus, 2.5 - 10 mg/day. |
| Efficacy assessments | At every quarterly visit, the investigator is required to confirm that the patient continues to have clinical benefit and may continue receiving study treatment. |
| Safety assessments | All adverse events and serious adverse events will be collected continuously throughout the study. |
| Other assessments | Not applicable. |
| Data analysis | Proportion of patients with clinical benefit as assessed by the investigator will be summarized at scheduled visits. The assessment of safety will be based mainly on the frequency of AEs and SAEs. |
| Key words | Everolimus roll-over study to better characterize the long term-term safety of everolimus in patients receiving everolimus in a Novartis-sponsored OGD&GMA study which has reached its objectives and who are benefiting from treatment with everolimus. |

# 1 Background

# 1.1 Overview of disease pathogenesis, epidemiology and current treatment

The roll-over study is designed to accept patients with varied disease origins. Please refer to the parent protocol for the disease background information and rationale for use of everolimus in their individual indications. See Section 1.2.1.2.

# 1.2 Introduction to investigational treatment(s) and other study treatment(s)

### 1.2.1 Overview of everolimus

Everolimus is a signal transduction inhibitor (STI) targeting mTOR, or more specifically, mTORC1 (mammalian 'target of rapamycin' complex 1). mTOR is a key serine-threonine kinase playing a central role in the regulation of cell growth, proliferation and survival. The regulation of mTORC1 signaling is complex, being modulated by mitogens, growth factors, energy and nutrient availability. mTORC1 is an essential regulator of global protein synthesis downstream on the PI3K/AKT/mTOR pathway, which is dysregulated in the majority of human cancers (Boulay and Lane 2007). Consistent with the known activity of mTORC1, its inhibition by everolimus has been shown to reduce cell proliferation, glycolysis and angiogenesis in solid tumors *in vivo*, both through direct antitumor cell activity and inhibition of the tumor stromal compartment.

mTOR is a key regulatory protein affecting various cell functions (Boulay and Lane 2007). The main known functions of mTOR include:

- Function as a sensor of mitogens, growth factors, energy and nutrient levels, facilitating cell-cycle progression through the G1 to- S- phase in appropriate growth conditions.
- Regulation of protein synthesis important for tumor cell proliferation and angiogenesis through inactivating eukaryotic initiation factor 4E binding proteins and activating the 40S ribosomal S6 kinases (e.g. p70S6K1). For example, activation of the mTOR pathway leads to:
  - Increased production of pro-angiogenic factors (e.g. VEGF) in tumors.
  - Tumor, endothelial and smooth muscle cell growth and proliferation.

# 1.2.1.1 Non-clinical experience

For latest information on the pre-clinical pharmacology and toxicology of everolimus please refer to the current Investigator Brochure (IB).

### 1.2.1.2 Clinical experience

In oncology, everolimus has been in clinical development since 2002 for patients with various hematologic and non-hematologic malignancies; as a single agent or in combination with antitumor agents. Malignancies that are currently being evaluated in Novartis sponsored

studies include the following: metastatic renal cell carcinoma (mRCC), breast cancer, pancreatic neuroendocrine tumors (pNET/NET), diffuse large B cell lymphoma (DLBCL), and hepatocellular cancer (HCC). In addition, treatment of patients with tuberous sclerosis complex (TSC) associated subependymal giant cell astrocytoma (SEGA), renal angiomyolipoma, and epilepsy are also being evaluated.

Phase I dose escalating studies, exploratory Phase I/II/III studies with everolimus as single agent or in combination with other anti-cancer agents, Phase II/III studies of everolimus in different indications, Phase III double-blind studies and Phase IV studies are contributing to the extensive clinical database.

Approximately 27,399 patients, (excluding those patients who received marketed Afinitor®/Votubia®, those on planned and roll over studies as well as excluding investigator-sponsored studies) have been enrolled in studies with everolimus as of 31-Mar-2015.

# Oncology

Everolimus was approved by FDA on 30-Mar-2009 under the trade name Afinitor<sup>®</sup> for the treatment of patients with advanced RCC after failure of treatment with sunitinib or sorafenib. The European Commission (EC) approved Afinitor<sup>®</sup> on 03-Aug-2009 for the treatment of patients with advanced RCC, whose disease has progressed on or after treatment with vascular endothelial growth factor (VEGF)-targeted therapy. As of 31-Mar-2015, Afinitor<sup>®</sup> has been approved in 121 countries worldwide for the treatment of patients with advanced RCC.

On 05-May-2011, FDA approved Afinitor® for the "treatment of progressive pNET in patients with unresectable, locally advanced or metastatic disease. Afinitor is not indicated for the treatment of patients with functional carcinoid tumors". The EC approved Afinitor® on 24-Aug-2011 for the treatment of unresectable or metastatic, well- or moderately-differentiated neuroendocrine tumors of pancreatic origin in adults with progressive disease. As of 31-Mar-2015, Afinitor® has been approved in >115 countries worldwide for the treatment of patients with pNET/neuroendocrine tumors.

On 20-Jul-2012, FDA approved Afinitor® for the treatment of postmenopausal women with advanced hormone receptor-positive, HER2-negative breast cancer in combination with exemestane, after failure of treatment with letrozole or anastrozole. The EC approved Afinitor® on 23-Jul-2012 for the treatment of hormone receptor-positive, HER2/neu negative advanced breast cancer, in combination with exemestane, in postmenopausal women without symptomatic visceral disease after recurrence or progression following a non-steroidal aromatase inhibitor. As of 31-Mar-2015, Afinitor® has been approved in >115 countries for the treatment of patients with advanced hormone receptor-positive, HER2-negative breast cancer.

# **Tuberous sclerosis complex**

Afinitor® received accelerated approval from FDA on 29-Oct-2010 for the "treatment of patients with SEGA associated with tuberous sclerosis complex (TSC) who require therapeutic intervention but are not candidates for curative surgical resection. The EC granted conditional approval on 02-Sep-2011 for everolimus under the trade name Votubia® for the "treatment of patients aged 3 years and older with SEGA associated with TSC who require

Page 15

therapeutic intervention but are not amenable to surgery. Afinitor® received accelerated approval from FDA on 26-Apr-2012 for the "treatment of adult patients with renal angiomyolipoma and TSC, not requiring immediate surgery

For further details please refer to the current everolimus IB.

### **Pharmacokinetics**

Everolimus is rapidly absorbed after oral administration, with a median time to peak blood levels ( $t_{max}$ ) of 1-2 hours postdose. The extent of absorption is estimated at above 11%. The area under the blood concentration-time curve (AUC) is dose-proportional over the dose range of 5 to 70 mg tested while maximum blood concentration  $C_{max}$  appears to plateau at dose levels higher than 20 mg. The terminal half-life in cancer patients averaged 30 hours, which is similar to that in healthy subjects. A high-fat meal altered the absorption of everolimus with 1.3 hour delay in  $t_{max}$ , a 60% reduction in  $C_{max}$  and a 16% reduction in AUC. In whole blood, approximately 80% of everolimus is contained in red blood cells. Of the fraction of drug contained in plasma, 74% is protein-bound. The apparent distribution volume (Vz/F) after a single dose was 4.7 L/kg. Everolimus is eliminated by metabolism, mainly by hydroxylation, then excreted into the feces >80%.

Everolimus is mainly metabolized by CYP3A4 in the liver and to some extent in the intestinal wall. Everolimus is also a substrate of P-glycoprotein (PgP). Therefore, absorption and subsequent elimination of systematically absorbed everolimus may be influenced by medicinal products that interact with CYP3A4 and/or P-glycoprotein. In vitro studies showed that everolimus is a competitive inhibitor of CYP3A4 and of CYP2D6 substrates, potentially increasing the concentrations of medicinal products eliminated by these enzymes. In two phase III clinical trials in patients following kidney transplantation, strong inhibitors of CYP3A4 (azoles, antifungals, cyclosporine, erythromycin) have been shown to reduce the clearance of everolimus therapy thereby increasing everolimus blood levels. Similarly, Rifampin, a strong inducer of CYP3A4, increases the clearance of everolimus thereby reducing everolimus blood levels. Another drug-drug interaction study of everolimus administered with a sensitive CYP3A4 substrate midazolam showed that while everolimus did not influence the hepatic metabolism of midazolam, it led to minor increases in bioavailability of midazolam likely due to influences of pre-systemic metabolism. Caution should be exercised when co-administering everolimus with CYP3A4 inhibitors, inducers, or substrates with a narrow therapeutic index.

# Pharmacodynamic studies

Pharmacokinetic/pharmacodynamic modeling based on inhibition in a peripheral biomarker (S6 kinase inhibition in peripheral blood mononuclear cells) suggests that 5 to 10 mg daily should be an adequate dose to produce a high-degree of sustained target inhibition. Furthermore, molecular pharmacodynamic (MPD) studies using IHC in biopsied tumor tissue assessed the degree of inhibition and its duration (for p-S6, p-4E-BP1 and p-Akt expression) with the daily and weekly dosing. The pathologist was blinded for the biopsy sequence. There was almost complete inhibition of p-S6 at all doses and schedules studied (p=0.001). Preliminary results suggest a dose-related decrease in p-4E-BP1 and increase in p-Akt expression with maximal effect at 10 mg daily and ≥50 mg weekly.

For further details please refer to the current everolimus IB.

### 2 Rationale

# 2.1 Study rationale and purpose

The purpose of this study is to better characterize the long-term safety of everolimus in patients who are currently receiving everolimus treatment in a Novartis-sponsored, OGD&GMA study that has reached its study objectives and are not progressing on the current study treatment as judged by the investigator. Parent studies eligible to participate in the roll-over study will be decided by Novartis. Investigator initiated trials (IITs) will not be included. The primary objective of the parent study must have been reached and the parent study must be in the process of being completed and reported.

Patients will continue to receive everolimus until one of the following occurs: no treatment benefit (disease progression) as judged by the investigator, unacceptable toxicity develops, consent withdrawal, protocol non-compliance, the investigator feels it is no longer in the patient's best interest to continue therapy, or the patient's death.

The roll-over protocol is designed to provide continued treatment with everolimus monotherapy to patients. If patients are receiving treatment of everolimus in combination with other approved therapies, they can participate in the roll-over study, but it is not intended for combination with unapproved or experimental treatments. Therefore, patients may be allowed to continue combination therapy with Sandostatin LAR® Depot if they are currently receiving this combination therapy on the parent protocol and at the discretion of the investigator. Sandostatin LAR® Depot is a formulation of octreotide which can be administered on a once monthly schedule and is available commercially worldwide.

Sandostatin LAR® Depot has been used to treat the symptoms associated with metastatic carcinoid tumors (flushing and diarrhea), and vasoactive intestinal peptide (VIP) secreting adenomas (watery diarrhea). For additional details please refer to the national prescribing information.

# 2.2 Rationale for the study design

This is a multi-center, open-label, phase IV study to better characterize the long-term safety of everolimus in patients being treated in a current Novartis-sponsored, OGD&GMA study and who are benefiting from treatment with everolimus. Patients may be allowed to continue combination therapy with Sandostatin LAR® Depot if they are currently receiving this combination therapy on the parent protocol and at the discretion of the investigator.

This study will not include a screening phase as patients will transfer directly from the parent study and will commence with everolimus as soon as they are consented and meet the inclusion criteria of the roll-over protocol.

# 2.3 Rationale for dose and regimen selection

Everolimus will be provided as 2.5 mg, 5 mg or 10 mg tablets. At the time of transition to the roll-over study, the starting dose of everolimus should be the same as the last dose that was

given in the parent study. Dose modification thereafter may be done at the discretion of the investigator based upon what is in the patient's best interest.

The roll-over protocol is designed to provide continued treatment with everolimus monotherapy to patients. If patients are receiving treatment of everolimus in combination with other approved therapies, they can participate in the roll-over study but it is not intended for combination with unapproved or experimental treatments. Therefore, for patients receiving everolimus in combination with Sandostatin LAR® Depot, Sandostatin LAR® Depot will be provided by Novartis or by the investigational site considering local regulations. At the time of transition to the roll-over study, the starting dose of Sandostatin LAR® Depot should be the same as the last dose that was given in the parent study.

# 2.4 Rationale for choice of combination drugs

Patients may be allowed to continue combination therapy with everolimus and Sandostatin LAR® Depot at the discretion of the investigator if they are currently receiving this combination therapy on the parent protocol and are deriving benefit as defined in the criteria of the parent protocol.

# 2.5 Rationale for choice of comparators drugs

Not applicable.

### 2.6 Risks & Benefits

# Postmenopausal women with hormone receptor-positive advanced breast cancer in combination with aromatase inhibitors, after prior endocrine therapy

Overall, everolimus + exemestane is considered to have a positive benefit-risk profile for postmenopausal women with hormone receptor-positive advanced breast cancer in combination with an aromatase inhibitor, after prior endocrine therapy; the benefits of therapy with everolimus + exemestane outweigh any potential risks.

# Advanced neuroendocrine tumors of pancreatic origin

Everolimus has a positive benefit-risk profile for patients with advanced pancreatic neuroendocrine tumors (pNET). Prior study results support the use of everolimus for the treatment of patients with advanced pNET. Results provided evidence that everolimus, in combination with octreotide depot, improved PFS in patients with advanced carcinoid tumors. The primary endpoint of the study was not met. More data is needed to better assess the benefit-risk of everolimus in this patient population.

# Renal cell carcinoma (RCC) after failure of treatment with sunitinib or sorafenib

Overall, everolimus is considered to have a positive benefit-risk profile for patients with advanced renal cell carcinoma after treatment failure with sunitinib or sorafenib. The benefits of therapy with everolimus outweigh any potential risks.

# 3 Objectives and endpoints

Objectives and related endpoints are described in Table 3-1 below.

# Table 3-1 Objectives and related endpoints

| Objective | Endpoint | Analysis |
|---|---|---|
| Primary | | |
| To evaluate long term safety data | Frequency and severity of AEs/SAEs | Refer to Section 10.4 |
| Secondary | | |
| To evaluate clinical benefit as assessed by the investigator | Proportion of patients with clinical benefit as assessed by the investigator at scheduled visits | Refer to Section 10.5 |

# 4 Study design

# 4.1 Description of study design

This is a multi-center, open label study to better characterize the long-term safety of everolimus in patients currently being treated in a Novartis-sponsored OGD&GMA study and who are not progressing on the current study treatment as judged by the investigator. Parent studies eligible to participate in the roll-over study will be decided by Novartis. Investigator initiated trials (IIT) will not be included.

There will be no screening period for this study. Eligible patients can start their treatment with everolimus as soon as they enter the study. All patients must report to the study site for their first visit and commence study participation. At that time, a quarterly supply of everolimus may be dispensed to the patient/or as per local practice.

Patients must return to the study center at least on a quarterly basis ( $\pm$  1 week) for resupply of study medication. Drug dispensing information and adverse events will be collected. The patient may return to the clinic at any given time as per standard of care or treating physician recommendation; however only the quarterly study visits will be recorded. Study medication dispensed will be recorded on the dose administration page.

All reported adverse events and serious adverse events will be collected throughout the study.

Patients will continue to be treated in the roll-over protocol until they are no longer benefiting from their everolimus treatment as judged by the investigator (disease progression), they develop unacceptable toxicities, they withdraw consent, they are non-compliant to the protocol, the investigator feels it is no longer in the patient's best interest to continue everolimus therapy or the patient dies, whichever comes first. At every quarterly visit, the investigator is required to confirm that the patient continues to have clinical benefit and may continue receiving study treatment.

A patient will reach the end of study when everolimus treatment is permanently discontinued.

The study is expected to remain open for 10 years or until such time that enrolled patients no longer need treatment with everolimus or are able to obtain commercial supply according to local regulations for their medical condition.

Figure 4-1 Study design

Parent Novartis Oncology CD&MA study: Everolimus

(tolerable effective dose)

Roll-over study:

\*Everolimus
(at assigned dose)

End of roll-over study:

Everolimus is permanently discontinued

<sup>\*</sup>Note: The starting everolimus (and Sandostatin LAR® Depot, if applicable) dose will be the same as the last dose received in the parent study.

# 4.2 Timing of interim analyses and design adaptations

Not applicable.

# 4.3 Definition of end of study

End of study is defined as either 10 years duration or when all patients on this study have permanently discontinued everolimus treatment and the end of treatment visit has been performed for each patient, whichever comes earlier.

# 4.4 Early study termination

The study is expected to remain open for 10 years or until such time that enrolled patients no longer need treatment with everolimus or are able to obtain commercial supply according to local regulations for their medical condition.

The study can be terminated at any time for any reason by Novartis. Should this be necessary, the prematurely withdrawn patient should be seen as soon as possible. The investigator may be informed of additional procedures to be followed in order to ensure that adequate consideration is given to the protection of the patient's interests. The investigator will be responsible for informing IRBs and/or ECs of the early termination of the trial.

# 5 Population

# 5.1 Patient population

The investigator or designee must ensure that only patients who meet all the following inclusion and none of the exclusion criteria are offered treatment in the study.

### 5.2 Inclusion criteria

Patients eligible for inclusion in this study have to meet all of the following criteria:

- 1. Patient is currently enrolled in a Novartis-sponsored, Oncology Global Development & Global Medical Affairs (OGD&GMA) study receiving everolimus or everolimus plus Sandostatin LAR® Depot and has fulfilled all their requirements in the parent study.
- 2. Patient is currently benefiting from the treatment with everolimus, as determined by the guidelines of the parent protocol.
- 3. Patient has demonstrated compliance, as assessed by the investigator, with the parent study protocol requirements.
- 4. Willingness and ability to comply with scheduled visits and treatment plans.
- 5. Written informed consent obtained prior to enrolling into the roll-over study.
  - If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.

### 5.3 Exclusion criteria

Patients eligible for this study must not meet any of the following criteria:

- 1. Patient has been permanently discontinued from everolimus study treatment in the parent study.
- 2. Patients who are receiving everolimus in combination with unapproved or experimental treatments.
- 3. Sexually active males, unless they use a condom during intercourse while taking drug and for 8 weeks after stopping study medication. Males also should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
- 4. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
- 5. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, **unless** they are using highly effective methods of contraception during dosing and for 8 weeks after stopping study treatment.
  - Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential

### **Highly effective** contraception methods include:

- Total abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
- Female Sterilization: Have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
- Male partner sterilization (at least 6 months prior to enrolling). [For female study subjects, the vasectomized male partner should be the sole partner for that patient]
- Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
- In case of use of oral contraception, women should have been stable on the same pill before taking study treatment.

If a study patient becomes pregnant or suspects being pregnant during the study or within 30 days after the final dose of everolimus, the investigator needs to be informed immediately and ongoing study treatment with everolimus has to be stopped immediately.

### 6 Treatment

# 6.1 Study treatment

Study treatment and investigational treatment refer to everolimus.

# 6.1.1 Dosing regimen

Table 6-1 Dose and treatment schedule

| Study treatments | Pharmaceutical form and route of administration | Dose | Frequency and/or Regimen |
|---|---|---|---|
| RAD001/everolimus | Tablet for oral use | 2.5 - 10 mg/day | Daily |

Everolimus will be provided as 2.5 mg, 5 mg or 10 mg tablets. The investigational treatment is to be stored in a secure locked area while under the responsibility of the investigator. Receipt and dispensing of investigational treatment must be recorded by an authorized person at the investigator's site. Everolimus for the roll-over study can be provided as local commercial material or global supply where appropriate.

At the time of transition to the roll-over study, the starting dose of everolimus should be the same as the last dose that was given in the parent study. Dose modification thereafter may be done at the discretion of the investigator based upon what is in the patient's best interest.

Patients will be instructed to take everolimus orally with a glass of water, once daily at the same time each day, either consistently with food or consistently without food. Dietary habits at the time of enrolling in the study from the parent study should be kept as consistent as possible throughout the study. The tablet should be swallowed as a whole and should not be chewed or crushed

Please refer to the current everolimus IB and Section 6.3 for further important information on potential dosing precautions regarding concomitant medication interaction with cytochrome p450, p-glycoprotein, and CYP3A4 and the recommended dosing guidance.

# 6.1.1.1 Dosing regimen for combination therapy treatment

The roll-over protocol is designed to provide continued treatment with everolimus monotherapy to patients. If patients are receiving treatment of everolimus in combination with other approved therapies, they can participate in the roll-over study, but it is not intended for combination with unapproved or experimental treatments. Therefore, for patients receiving everolimus in combination with Sandostatin LAR® Depot on the parent protocol, Sandostatin LAR® Depot will continue to be provided by Novartis or by the investigational site considering local regulations. At the time of transition to the roll-over study, the starting dose of Sandostatin LAR® Depot should be the same as the last dose that was given in the parent study.

Table 6-2 Combination therapy dose and treatment schedule

| Study treatments | Pharmaceutical form<br>and route of<br>administration | Dose | Frequency and/or<br>Regimen |
|---|---|---|---|
| Sandostatin LAR® (if applicable) | Intramuscular injection | At discretion of treating physician | At discretion of treating physician |

# 6.1.2 Ancillary treatments

Not applicable.

### 6.1.3 Rescue medication

Not applicable.

### 6.1.4 Guidelines for continuation of treatment

The starting dose of everolimus should be the same as the last dose that was given in the parent everolimus study. Following the starting dose, patient's may have their dose of everolimus (2.5-10 mg/day) adjusted based on the investigator's judgment of what dose is in the patient's best interest.

### 6.1.5 Treatment duration

Patients will continue to be treated in the roll-over protocol until they are no longer benefiting from their everolimus treatment as judged by the investigator (disease progression), they develop unacceptable toxicities, they withdraw consent, they are non-compliant to the protocol, the investigator feels it is no longer in the patient's best interest to continue everolimus therapy or the patient dies, whichever comes first. At every quarterly visit the investigator is required to confirm that the patient continues to have clinical benefit and may continue receiving study treatment. A patient will reach the end of the roll-over study when everolimus treatment is permanently discontinued.

The study is expected to remain open for 10 years or until such time that enrolled patients no longer need treatment with everolimus or are able to obtain commercial supply according to local regulations for their medical condition.

# 6.2 Dose escalation guidelines

Not applicable.

### 6.3 Dose modifications

# 6.3.1 Dose modification and dose delay

Patients will begin the roll-over study at the same dose as the last dose administered in the parent protocol. Dose adjustments are permitted to allow the patient to continue the study treatment at the investigator's discretion. Dose modifications may be applied at the investigator's discretion in conjunction with the most current IB.

Everolimus and Sandostatin LAR Depot® dose changes must be recorded on the Dosage Administration Record eCRFs.

# 6.3.2 Follow-up for toxicities

Patients whose treatment is interrupted or permanently discontinued due to an adverse event or clinically significant laboratory value, should be followed up at least once a week (or more frequently if clinically indicated) for 4 weeks, and subsequently at approximately 4-week intervals, until resolution or stabilization of the event, whichever comes first.

Appropriate clinical experts such as ophthalmologist, endocrinologist, dermatologist, psychiatrists etc. should be consulted as deemed necessary. Patients must be followed for adverse events and serious adverse events for 30 days following the last dose of everolimus.

## 6.3.2.1 Follow up on potential drug-induced liver injury (DILI) cases

Patients with transaminase increase combined with TBIL increase may be indicative of potential DILI, and should be considered as clinically important events.

The threshold for potential DILI may depend on the patient's baseline AST/ALT and TBIL value; patients meeting any of the following criteria will require further follow-up as outlined below:

- For patients with normal ALT and AST and TBIL value at baseline: AST or ALT > 3.0 x ULN combined with TBIL > 2.0 x ULN
- For patients with elevated AST or ALT or TBIL value at baseline: [AST or ALT > 2 x baseline AND > 3.0 x ULN] OR [AST or ALT > 8.0 x ULN], combined with [TBIL > 2 x baseline AND > 2.0 x ULN]

Medical review needs to ensure that liver test elevations are not caused by cholestasis, defined as ALP elevation > 2.0 x ULN with R value < 2 in patients without bone metastasis, or elevation of ALP liver fraction in patients with bone metastasis.

Note: (The R value is calculated by dividing the ALT by the ALP, using multiples of the ULN for both values. It denotes whether the relative pattern of ALT and/or ALP elevation is due to cholestatic ( $R \le 2$ ), hepatocellular ( $R \ge 5$ ), or mixed ( $R \ge 2$  and  $R \ge 1$ ) liver injury).

In the absence of cholestasis, these patients should be immediately discontinued from study drug treatment, and repeat LFT testing as soon as possible, preferably within 48 hours from the awareness of the abnormal results. The evaluation should include laboratory tests, detailed history, physical assessment and the possibility of liver metastasis or new liver lesions, obstructions/compressions, etc.

- 1. Laboratory tests should include ALT, AST, albumin, creatine kinase, total bilirubin, direct and indirect bilirubin, GGT, prothrombin time (PT)/INR and alkaline phosphatase.
- 2. A detailed history, including relevant information, such as review of ethanol, concomitant medications, herbal remedies, supplement consumption, history of any pre-existing liver conditions or risk factors, should be collected.
- 3. Further testing for acute hepatitis A, B, C or E infection and liver imaging (e.g. biliary tract) may be warranted.
- 4. Obtain PK sample, as close as possible to last dose of study drug, if PK analysis is performed in the study.

5. Additional testing for other hepatotropic viral infection (CMV, EBV or HSV), autoimmune hepatitis or liver biopsy may be considered as clinically indicated or after consultation with specialist/hepatologist.

All cases confirmed on repeat testing meeting the laboratory criteria defined above, with no other alternative cause for LFT abnormalities identified should be considered as "medically significant", thus, met the definition of SAE (Section 8.2.1) and reported as SAE using the term "potential drug-induced liver injury". All events should be followed up with the outcome clearly documented.

# 6.3.3 Anticipated risks and safety concerns of the study drug

It is anticipated that the patients entering the roll-over protocol have tolerated everolimus treatment and are anticipated to benefit from continued treatment.

Guidelines and recommendations for the management of specific everolimus study drug induced toxicities (hyperglycemia, hyperlipidemia, stomatitis, infectious pneumonitis, reactivation of Hepatitis B and C) are provided in the current everolimus Investigator Brochure

### 6.4 Concomitant medications

# 6.4.1 Permitted concomitant therapy

In general, concomitant medications/therapies deemed necessary for the supportive care of the patient is permitted.

# 6.4.2 Permitted concomitant therapy requiring caution and/or action

Everolimus is metabolized by CYP3A4 in the liver and to some extent in the intestinal wall. Therefore, the following are recommended:

- Co-administration with strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, ritonavir) or P-glycoprotein (PgP) inhibitor should be avoided.
- Co-administration with moderate CYP3A4 inhibitors (e.g., erythromycin, fluconazole) or PgP inhibitors should be used with caution. If a patient requires co-administration of moderate CYP3A4 inhibitors or PgP inhibitors, reduce the dose of study drug to half the currently used dose. Additional dose reductions to every other day may be required to manage toxicities. If the inhibitor is discontinued, the study drug dose should be returned to the dose used prior to initiation of the moderate CYP3A4/PgP inhibitor.
- Seville orange, star fruit, grapefruit and their juices affect P450 and PgP activity. Concomitant use should be avoided.
- Co-administration with strong inducers of CYP3A4 should be avoided. If a patient requires co-administration of strong CYP3A4 inducers (i.e., phenytoin, carbamazepine, rifampin, rifabutin, phenobarbital, St. John's wort), an increase in the dose of study drug up to twice the currently used daily dose should be considered, 5mg increments. Enzyme induction usually occurs within 7-10 days; therefore study drug dose should be increased by one increment 7 days after the start of the inducer therapy. If no safety concerns are seen within the next 7 days, the dose can be increased again one additional increment up

to a maximum of twice the daily dose used prior to initiation of the strong CYP3A4 inducer.

 This dose adjustment of study drug is intended to achieve similar AUC to the range observed without inducers. However, there are no clinical data with this dose adjustment in patients receiving strong CYP3A4 inducers. If the strong inducer is discontinued the study drug dose should be returned to the dose used prior to initiation of the strong CYP3A4/PgP inducer.

Please refer to Table 6-3 listing relevant inducers and inhibitors of CYP3A and to Table 6-4 for a list of relevant substrates, inducers, and inhibitors of PgP. Please refer to the most recent Investigator's Brochure for a complete list.

# Table 6-3 Clinically relevant drug interactions: inducers, and inhibitors of isoenzyme CYP3A

### Inducers

### Strong inducers:

avasimibe, carbamazepine, mitotane, phenobarbital, phenytoin, rifabutin, rifampin (rifampicin), St. John's wort (hypericum perforatum)

### Moderate inducers:

bosentan, efavirenz, etravirine, genistein, modafinil, nafcillin, ritonavir, [talviraline], thioridazine, tipranavir

### Weak inducers

amprenavir, aprepitant, armodafinil (R-modafinil), bexarotene, clobazam, danshen, dexamethasone, Echinacea, garlic (allium sativum), gingko (ginkgo biloba), glycyrrhizin, methylprednisolone, nevirapine, oxcarbazepine, pioglitazone, prednisone, [pleconaril], primidone, raltegravir, rufinamide, sorafenib, telaprevir, terbinafine, topiramate, [troglitazone], vinblastine

### **Inhibitors**

### Strong inhibitors:

**boceprevir**, clarithromycin, cobicistat, conivaptan, elvitegravir, indinavir, itraconazole, ketoconazole, lopinavir, mibefradil, nefazodone, nelfinavir, posaconazole (Krishna et al 2009), ritonavir, saquinavir, **telaprevir**, telithromycin, tipranavir, troleandamycin, voriconazole

### Moderate inhibitors:

Amprenavir, aprepitant, atazanavir, casopitant, cimetidine, ciprofloxacin, cyclosporine, darunavir, diltiazem, dronedarone, erythromycin, fluconazole, fosamprenavir, grapefruit juice (citrus parasidi fruit juice), imatinib, schisandra sphenanthera, tofisopam, verapamil

# Table 6-4 Clinically relevant drug interactions: substrates, inducers, inhibitors of PgP and PgP/CYP3A dual inhibitors

### **Substrates**

colchicine, digoxin, fexofenadine, indinavir, paclitaxel, talinolol, topotecan, vincristine, everolimus

### Inducers

rifampin, St John's wort

### PgP Inhibitors and PgP/CYP3A Dual Inhibitors

amiodarone, azithromycin, captopril, carvedilol, clarithromycin, conivaptan, diltiazem, dronedarone, elacridar, erythromycin, felodipine, fexofenadine, fluvoxamine, ginkgo (ginkgo biloba), indinavir, itraconazole, lopinavir, mibefradil, milk thistle (silybum marianum), nelfinavir, nifedipine, nitrendipine, paroxetine, quercetin, quinidine, ranolazine, rifampin, ritonavir, saquinavir, Schisandra chinensis, St John's wort (hypericum perforatum), talinolol, Telaprevir, telmisartan, ticagrelor, tipranavir, tolvaptan, valspodar, verapamil

Reference: Internal Clinical Pharmacology Drug-drug interaction (DDI) memo, updated 29-Oct-2012 which summarizes DDI data from three sources including the FDA's "Guidance for Industry, Drug Interaction Studies", the University of Washington's Drug Interaction Database, and Indiana University School of Medicine's Drug Interaction Table.

### **Vaccinations**

The use of live vaccines and close contact with those who have received live vaccines should be avoided during treatment with everolimus. Examples of live vaccines are: intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid vaccines.

For further details refer to the current everolimus Investigator's Brochure.

# 6.4.3 Prohibited concomitant therapy

Treatment with systemic anticancer agents (chemotherapy, hormone therapy, targeted or biologic agents) other than everolimus is not permitted until disease progression is documented and everolimus is permanently discontinued.

### 6.4.4 Use of Bisphosphonates (or other concomitant agents)

Not applicable.

# 6.5 Patient numbering, treatment assignment or randomization

# 6.5.1 Patient numbering

Each patient is identified in the study by a Subject Number (Subject No.), that is assigned when the patient is first enrolled in the roll-over study and is retained as the primary identifier for the patient throughout his/her entire participation in the trial. The Subject No. consists of the Center Number (Center No.) (as assigned by Novartis to the investigative site) with a sequential patient number suffixed to it, so that each subject is numbered uniquely across the entire database. Upon signing the informed consent form, the patient is assigned to the next sequential Subject No. available to the investigator through the Oracle Clinical RDC interface (OCRDC).

Additionally an eCRF will be completed that identifies the patient by gender and date of birth and previous study, site/center and subject number.

# 6.5.2 Treatment assignment or randomization

All consented patients who meet all the inclusion criteria and none of the exclusion criteria are eligible to receive everolimus.

# 6.5.3 Treatment blinding

Not applicable.

# 6.6 Study drug preparation and dispensation

The investigator or responsible site personnel must instruct the patient or caregiver to take the study drugs as per protocol. Study drug(s) will be dispensed to the patient by authorized site personnel only. All everolimus dosages prescribed to the patient and all dose changes during the study must be recorded on the Everolimus Dosage Administration Record eCRF.

Table 6-5 Preparation and dispensing

| Study treatments | Dispensing | Preparation |
|---|---|---|
| Everolimus | Blister packed tablets (2.5 – 10 mg) including instructions for administration will be dispensed by study personnel on an outpatient basis. Patients will be provided with an adequate supply of study treatment for self-administration at home until at least their next scheduled quarterly (12 weeks ± 1 week) study visit. | Not applicable |
| | If study drug is supplied by Novartis Drug Supply Management, the supply may be dispensed more frequently if required based on local practice or drug expiration date. | |

## 6.6.1 Study treatment packaging and labeling

Everolimus for the roll-over study can be provided where appropriate as local commercial material or as global open-label supply, packed and labeled under the responsibility of Novartis Drug Supply Management. Study treatment labels will be in the local language and comply with the legal requirements of each country. They will include storage conditions for the drug but no information about the patient.

If everolimus is provided and labeled in-country, the locally-approved form and packaging of everolimus will be used.

Table 6-6 Packaging and labeling

| Study treatments | Packaging | Labeling (and dosing frequency) |
|---|---|---|
| Everolimus | Tablets in blisters* | As per local requirements |
| * For centrally supplied medication. If everolimus is sourced and labeled in-country/locally, the locally-approved | | |
| form, packaging and labeling of everolimus will be used. | | |

# 6.6.2 Drug supply and storage

Study treatments must be received by designated personnel at the study site, handled and stored safely and properly, and kept in a secured location to which only the investigator and designated site personnel have access. Upon receipt, everolimus should be stored according to the instructions specified on the drug labels and in the Investigator's Brochure.

Table 6-7 Supply and storage of study treatments

| Study treatments | Supply | Storage |
|---|---|---|
| Everolimus | Centrally or locally supplied by | Refer to study treatment label or local product |
| | Novartis | information |

# 6.6.3 Study drug compliance and accountability

# 6.6.3.1 Study drug compliance

Compliance will be assessed by the investigator and/or study personnel at each patient visit and information provided by the patient and/or caregiver will be captured in the Drug Accountability Form and other relevant source documents.

## 6.6.3.2 Study drug accountability

The investigator or designee must maintain an accurate record of the shipment and dispensing of study treatment in a drug accountability log. Drug accountability will be noted by the field monitor during site visits and at the completion of the study. Patients will be asked to return all unused study treatment and packaging on a regular basis, at the end of the study or at the time of study treatment discontinuation.

# 6.6.3.3 Handling of other study treatment

If the patient was receiving a combination therapy with an approved, commercially available treatment with everolimus in the parent protocol, and is eligible for the roll-over study, this combination therapy will be allowed until the patient permanently discontinues everolimus. All Sandostatin LAR® Depot dosages prescribed to the patient and all dose changes during the study must be recorded on the Sandostatin Dosage Administration Record eCRF.

Dispensation, compliance and accountability of any combination therapy administered to the patient is under the supervision and discretion of the investigator. Sandostatin LAR® Depot will be provided by Novartis or by the investigational site considering local regulations. Sandostatin LAR® Depot will be distributed in country-specific approved packaging.

# 6.6.4 Disposal and destruction

At study close-out, and, as appropriate during the course of the study, the investigator will return all used and unused study treatment, packaging, drug labels, and a copy of the completed drug accountability log to the Novartis monitor or to the Novartis address provided in the investigator folder at each site.

The study drug can only be destroyed once the study drug accountability check has been done by the monitor. The study drug can be destroyed at the local Novartis facility or by a third party, as appropriate.

# 7 Visit schedule and assessments

# 7.1 Study flow and visit schedule

Table 7-1 lists all of the assessments and indicates with an "X", the visits when they are performed. A visit window of  $\pm$  1 week is allowed. All data obtained from these assessments must be supported in the patient's source documentation.

The table indicates in the "Category" column which assessments produce data to be entered in the database (D) or documented at the site level in the source documents (S).

Table 7-1 Visit evaluation schedule

| | Category | Protocol<br>reference<br>section | Enrolment | Quarterly (every 12 weeks± 1 week) visits during treatment phase | End of treatment (EoT) | 30 day safety<br>follow-up post last<br>dose of study drug/<br>End of Study |
|---|---|---|---|---|---|---|
| Visit Number | | | 1 | Visit 2, 3, 4 etc. | 777 | |
| Obtain informed consent | D | 7.1.2 | Х | | | |
| Patient's previous study,site, and subject number | D | 7.1.2.3 | х | | | |
| Demography | D | 7.1.2.3 | Х | | | |
| Relevant medical history/current medical conditions | D | 7.1.2.3 | х | | | |
| Inclusion/exclusion criteria | D | 5.2 / 5.3 | Х | | | |
| Serum pregnancy testing | D | 7.2.2 | Х | | Х | |
| Urine pregnancy testing | S/D | 7.2.2 | | monthly | | |
| Adverse events and Serious adverse events | D | 8.1 / 8.2 | х | continuous | х | х |
| Everolimus dosing administration | D | 6.6 | х | continuous | | |
| Sandostatin LAR® Depot dosing administration (if applicable) | D | 6.6 | x | continuous | | |
| Confirmation of Clinical Benefit from Study Treatment | D | 6.1.5 | х | continuous | | |
| End of study treatment | D | 7.1.5 | | | x | |
| Study evaluation completion | D | 7.1.5 | | | | Х |

# 7.1.1 Molecular pre-screening

Not applicable.

# 7.1.2 Screening

At the enrollment visit the patient will complete a written informed consent. There will be no screening period for this study. Once consented, patients will be evaluated for eligibility via the inclusion and exclusion criteria.

# 7.1.2.1 Eligibility screening

Not applicable.

# 7.1.2.2 Information to be collected on screening failures

Not applicable.

### 7.1.2.3 Patient demographics and other baseline characteristics

For patients that are eligible to participate in this roll-over study, the patients' gender, date of birth, previous study, site/center and subject number, and relevant medical history will be collected.

# 7.1.3 Run-in period

Not applicable.

### 7.1.4 Treatment period

The starting dose of everolimus on this roll-over protocol will be the same as the last dose that was given in the parent everolimus study. A 3 month supply of everolimus will be dispensed to the patient, or what is allowed according to local practice/regulations.

Patients must return to the study center on a quarterly basis (12 weeks  $\pm$  1 week) for resupply of study medication at which time drug dispensing information and adverse event information will be collected. At this time the dose of everolimus is based on the investigator's judgment. At every quarterly visit, the investigator is required to confirm that the patient continues to have clinical benefit and may continue treatment with study drug.

The study is expected to remain open for 10 years or until such time that enrolled patients no longer need treatment with everolimus or are able to obtain commercial supply according to local regulations for their medical condition.

# 7.1.5 Discontinuation of study treatment

Patients will continue to be treated until they are no longer benefiting from everolimus treatment, develop unacceptable toxicities, withdraw consent, are non-compliant to the protocol, or the patient dies, whichever comes first.

At the time the patient discontinues study treatment, a visit should be scheduled as soon as possible, at which time the End of Treatment visit will be performed. End of Treatment

information will be completed in the eCRF giving the date and reason for stopping the study treatment (see Section 7.1.5.1).

At a minimum, all patients who discontinue study treatment, including those who refuse to return for a final visit, will be contacted for the required safety evaluation during the 30 days following the last dose of study treatment. The completion of the Study Evaluation Completion eCRF page is required any time a patient discontinues from the study and must be completed 30 days after the end of treatment.

Patients who discontinue study treatment should be considered withdrawn from the study after the final visit assessments are performed or when it is clear that the patient will not return for these assessments.

If a study withdrawal occurs, or if the patient fails to return for visits, the investigator must determine the primary reason for a patient's withdrawal from the study and record this information on the appropriate eCRF page.

A patient will reach the end of study when everolimus treatment is permanently discontinued and there will be **no** further follow-up study visits.

### 7.1.5.1 Withdrawal of consent

Patients may voluntarily withdraw consent to participate in the study for any reason at any time. Withdrawal of consent occurs only when a patient does not want to participate in the study any longer, and does not want any further visits or assessments, and does not want any further study related contact.

Novartis will continue to retain and use all research results that have already been collected for the study evaluation. All biological samples that have already been collected may be retained and analyzed at a later date (or as required by local regulations).

If a patient withdraws consent, the investigator should make a reasonable effort (e.g. telephone, e-mail, letter) to understand the primary reason for this decision and record this information.

Everolimus must be discontinued and no further assessments conducted.

Further attempts to contact the patient are not allowed unless safety findings require communication or follow up.

Patients may be withdrawn from the study if any of the following occur:

- 1. Adverse event(s).
- 2. Subject withdrew consent.
- 3. Lost to follow-up.
- 4. Administrative problems.
- 5. Death.
- 6. Disease progression.
- 7. Treatment duration completed as per protocol.
- 8. Protocol deviation
- 9. Sponsor decision

# 7.1.5.2 Replacement policy

Not applicable.

# 7.1.6 Follow up for safety evaluations

All patients must be followed up for safety evaluations for 30 days after the last dose of everolimus. At the end of this period, the investigator should contact the patient to inquire about any adverse events or serious adverse events observed during this period. This could be done via a phone contact. Following this there are **no** further follow-up study visits.

### 7.1.7 Lost to follow-up

For patients whose status is unclear because they fail to appear for study visits without stating an intention to withdraw consent, the investigator should show "due diligence" by contacting the patient, family or family physician as agreed in the informed consent and by documenting in the source documents steps taken to contact the patient, e.g. dates of telephone calls, registered letters, etc. A patient should not be considered lost to follow-up until due diligence has been completed. Patients lost to follow up should be recorded as such on the appropriate Disposition CRF.

# 7.2 Assessment types

# 7.2.1 Efficacy assessments

At every quarterly visit, the investigator is required to confirm that the patient continues to have clinical benefit and may continue receiving study treatment.

# 7.2.2 Safety and tolerability assessments

Safety will be monitored by collecting Adverse Events throughout the study on a continuous basis. See Section 8.

Women of child-bearing potential must complete the following pregnancy tests:

- Baseline/Enrollment serum pregnancy test done locally
- Every 4 weeks during treatment urine pregnancy test. Can be administered at patient's home.
- End of Treatment visit serum pregnancy test done locally

Women of child-bearing potential who administer urine pregnancy testing at home should complete a simple diary with the dates and the outcome of the urine pregnancy test while on study treatment. In case of a positive pregnancy test, the instructions in Section 8.4 should be followed.

### 7.2.3 Pharmacokinetics

Not applicable.

### 7.2.4 Biomarkers

Not applicable.

### 7.2.5 Resource utilization

Not applicable.

# 7.2.6 Patient reported outcomes

Not applicable.

# 8 Safety monitoring and reporting

# 8.1 Adverse events

# 8.1.1 Definitions and reporting

An adverse event is defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occur after patient's signed informed consent has been obtained.

Adverse events of special interest as noted in Section 8.1.3 will be reported as serious adverse events.

Abnormal laboratory values or test results occurring after informed consent constitute adverse events only if they induce clinical signs or symptoms, are considered clinically significant, require therapy (e.g., hematologic abnormality that requires transfusion or hematological stem cell support), or require changes in study medication(s).

Any ongoing adverse events from the parent study will be captured as medical history in the roll-over database. Any AE that begins (or worsens) after signing of the informed consent for the rollover and during the 30-day (or 28-day) safety follow up period defined in the parent protocol should be reported in both clinical databases.

Adverse event monitoring should be continued for at least 30 following the last dose of study treatment. Adverse events (including lab abnormalities that constitute AEs) should be described using a diagnosis whenever possible, rather than individual underlying signs and symptoms. When a clear diagnosis cannot be identified, each sign or symptom should be reported as a separate Adverse Event.

Adverse events will be assessed according to the current version of the Common Terminology Criteria for Adverse Events (CTCAE). If CTCAE grading does not exist for an adverse event, the severity of mild, moderate, severe, and life-threatening, corresponding to Grades 1 - 4, will be used. CTCAE Grade 5 (death) will not be used in this study; rather, information about deaths will be collected on the EOT page.

The occurrence of adverse events should be sought by non-directive questioning of the patient (subject) during the screening process after signing informed consent and at each visit during the study. Adverse events also may be detected when they are volunteered by the patient (subject) during the screening process or between visits, or through physical examination, laboratory test, or other assessments. As far as possible, each adverse event should be evaluated to determine:
- 1. The severity grade (CTCAE Grade 1-4)
- 2. Its duration (Start and end dates)
- 3. Its relationship to the study treatment (reasonable possibility that AE is related: No, Yes)
- 4. Action taken with respect to study or investigational treatment (none, dose adjusted, temporarily interrupted, permanently discontinued, unknown, not applicable)
- 5. Whether medication or therapy was given (no concomitant medication/non-drug therapy, concomitant medication/non-drug therapy)
- 6. Whether it is serious, where a serious adverse event (SAE) is defined as in Section 8.2.1

If the event worsens the event should be reported a second time in the CRF noting the start date when the event worsens in toxicity. For grade 3 and 4 adverse events only, if improvement to a lower grade is determined a new entry for this event should be reported in the CRF noting the start date when the event improved from having been Grade 3 or Grade 4.

All adverse events should be treated appropriately. If a concomitant medication or non-drug therapy is given, this action should be recorded on the Adverse Event CRF.

Once an adverse event is detected, it should be followed until its resolution or until it is judged to be permanent, and assessment should be made at each visit (or more frequently, if necessary) of any changes in severity, the suspected relationship to the study treatment, the interventions required to treat it, and the outcome.

Progression of malignancy (including fatal outcomes), if documented by use of appropriate method (for example, as per RECIST criteria for solid tumors or as per Cheson's guidelines for hematological malignancies), should not be reported as a serious adverse event.

Adverse events separate from the progression of malignancy (example, deep vein thrombosis at the time of progression or hemoptysis concurrent with finding of disease progression) will be reported as per usual guidelines used for such events with proper attribution regarding relatedness to the drug.

#### 8.1.2 Laboratory test abnormalities

#### 8.1.2.1 Definitions and reporting

Laboratory abnormalities that constitute an Adverse event in their own right (are considered clinically significant, induce clinical signs or symptoms, require concomitant therapy or require changes in study treatment), should be recorded on the Adverse Events CRF. Whenever possible, a diagnosis, rather than a symptom should be provided (e.g. anemia instead of low hemoglobin). Laboratory abnormalities that meet the criteria for Adverse Events should be followed until they have returned to normal or an adequate explanation of the abnormality is found. When an abnormal laboratory or test result corresponds to a sign/symptom of an already reported adverse event, it is not necessary to separately record the lab/test result as an additional event.

Laboratory abnormalities, that do not meet the definition of an adverse event, should not be reported as adverse events. A Grade 3 or 4 event (severe) as per CTCAE does not automatically indicate a SAE unless it meets the definition of serious as defined below and/or as per investigator's discretion. A dose hold or medication for the lab abnormality may be

required by the protocol in which case the lab abnormality would still, by definition, be an adverse event and must be reported as such.

#### 8.1.3 Adverse events of special interest

Adverse events of special interest (AESI) are defined as events (serious or non-serious) which are ones of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor may be appropriate. Such events may require further investigation in order to characterize and understand them.

Adverse events of special interest are defined on the basis of an ongoing review of the safety data. AESIs are discussed in detail in the Investigator Brochure.

In addition to all serious adverse events reported on a continuous basis throughout the study, the investigator should use the SAE form to report the following medically significant potential risks noted in the Novartis Risk Management Plan for everolimus:

- Development toxicity
- Reproductive (teratogenicity) toxicity
- Intestinal obstruction /ileus
- Male infertility
- Pancreatitis
- Cholelithiasis
- Muscle-wasting/Muscle-loss

#### 8.2 Serious adverse events

#### 8.2.1 Definitions

Serious adverse event (SAE) is defined as one of the following:

- Is fatal or life-threatening
- Results in persistent or significant disability/incapacity
- Constitutes a congenital anomaly/birth defect
- Is medically significant, i.e., defined as an event that jeopardizes the patient or may require medical or surgical intervention to prevent one of the outcomes listed above
- Requires inpatient hospitalization or prolongation of existing hospitalization,
- Note that hospitalizations for the following reasons should not be reported as serious adverse events:
  - Routine treatment or monitoring of the studied indication, not associated with any deterioration in condition
  - Elective or pre-planned treatment for a pre-existing condition that is unrelated to the indication under study and has not worsened since signing the informed consent
  - Social reasons and respite care in the absence of any deterioration in the patient's general condition

Protocol No. CRAD001C2X01B

• Note that treatment on an emergency outpatient basis that does not result in hospital admission and involves an event not fulfilling any of the definitions of a SAE given above is not a serious adverse event

#### 8.2.2 Reporting

To ensure patient safety, every SAE, regardless of suspected causality, occurring after the patient has provided informed consent and until at least 30 days after the patient has stopped study treatment must be reported to Novartis within 24 hours of learning of its occurrence.

Any SAE that begins or worsens after signing of the informed consent for the roll-over and during the 30-day (or 28-day) safety follow up period defined in the parent protocol should be reported as an adverse event in both clinical databases; however, only one SAE report will be sent to Novartis.

- Any SAE that begins or worsens **during** the 30-day (or 28-day) safety follow up period specified in the parent study, should have an SAE report submitted to Novartis with the parent protocol study number.
- Any SAE that begins or worsens **after** the 30-day (or 28-day) safety follow-up period specified in the parent study, should have an SAE report submitted to Novartis with the roll-over protocol study number.

Any additional information for the SAE including complications, progression of the initial SAE, and recurrent episodes must be reported as follow-up to the original episode within 24 hours of the investigator receiving the follow-up information. An SAE occurring at a different time interval or otherwise considered completely unrelated to a previously reported one should be reported separately as a new event.

It is important to use the right SAE form with the correct protocol number for these two scenarios, to avoid confusion in SAE processing. For a patient already on the roll-over protocol but follow up information is reported for the previous SAEs in the parent protocol, it must be clearly labeled that this is for the parent protocol number.

Any SAEs experienced after the 30 day safety evaluation follow-up period should only be reported to Novartis if the investigator suspects a causal relationship to the study treatment.

Information about all SAEs is collected and recorded on the Serious Adverse Event Report Form; all applicable sections of the form must be completed in order to provide a clinically thorough report. The investigator must assess and record the relationship of each SAE to each specific study treatment (if there is more than one study treatment), complete the SAE Report Form in English, and submit the completed form within 24 hours to Novartis. Detailed instructions regarding the SAE submission process and requirements for signatures are to be found in the investigator folder provided to each site.

Follow-up information is submitted in the same way as the original SAE Report. Each reoccurrence, complication, or progression of the original event should be reported as a followup to that event regardless of when it occurs. The follow-up information should describe whether the event has resolved or continues, if and how it was treated, whether the blind was broken or not, and whether the patient continued or withdrew from study participation. If the SAE is not previously documented in the Investigator's Brochure or Package Insert (new occurrence) and is thought to be related to the Novartis study treatment, an oncology Novartis Drug Safety and Epidemiology (DS&E) department associate may urgently require further information from the investigator for Health Authority reporting. Novartis may need to issue an Investigator Notification (IN), to inform all investigators involved in any study with the same drug that this SAE has been reported. Suspected Unexpected Serious Adverse Reactions (SUSARs) will be collected and reported to the competent authorities and relevant ethics committees in accordance with Directive 2001/20/EC or as per national regulatory requirements in participating countries.

## 8.3 Emergency unblinding of treatment assignment

Not applicable.

#### 8.4 Pregnancies

To ensure patient safety, each pregnancy occurring while the patient is on study treatment must be reported to Novartis within 24 hours of learning of its occurrence. The pregnancy should be followed up to determine outcome, including spontaneous or voluntary termination, details of the birth, and the presence or absence of any birth defects, congenital abnormalities, or maternal and/or newborn complications.

Pregnancy should be recorded on a Clinical Trial Pregnancy Form and reported by the investigator to the oncology Novartis Drug Safety and Epidemiology Department (DS&E). Pregnancy follow-up should be recorded on the same form and should include an assessment of the possible relationship to the study treatment of any pregnancy outcome. Any SAE experienced during pregnancy must be reported on the SAE Report Form.

Pregnancy outcomes must be collected for the female partners of any males who took study treatment in this study. Consent to report information regarding these pregnancy outcomes should be obtained from the mother.

Preclinical data regarding reproductive toxicity is described in the most recent Investigator Brochure. The potential reproductive risk for humans is unknown. Women of childbearing potential should be advised to use highly effective contraception methods while they are receiving everolimus and up to 8 weeks after treatment has been stopped. If a pregnancy occurs while on study treatment, the newborn will be followed for at least 12 months.

# 8.5 Warnings and precautions

No evidence available at the time of the approval of this study protocol indicated that special warnings or precautions were appropriate, other than those noted in the provided Investigator Brochure. Additional safety information collected between IB updates will be communicated in the form of Investigator Notifications. This information will be included in the patient informed consent and should be discussed with the patient during the study as needed.

# 8.6 Data Monitoring Committee

Not applicable.

## 8.7 Steering Committee

Not applicable.

## 9 Data collection and management

## 9.1 Data confidentiality

Information about study subjects will be kept confidential and managed under the applicable laws and regulations. Those regulations require a signed subject authorization informing the subject of the following:

- What protected health information (PHI) will be collected from subjects in this study
- Who will have access to that information and why
- Who will use or disclose that information
- The rights of a research subject to revoke their authorization for use of their PHI.

In the event that a subject revokes authorization to collect or use PHI, the investigator, by regulation, retains the ability to use all information collected prior to the revocation of subject authorization. For subjects that have revoked authorization to collect or use PHI, attempts should be made to obtain permission to collect follow-up safety information (e.g. has the subject experienced any new or worsened AEs) at the end of their scheduled study period.

The data collection system for this study uses built-in security features to encrypt all data for transmission in both directions, preventing unauthorized access to confidential participant information. Access to the system will be controlled by a sequence of individually assigned user identification codes and passwords, made available only to authorized personnel who have completed prerequisite training.

# 9.2 Site monitoring

Before study initiation, at a site initiation visit or at an investigator's meeting, Novartis personnel (or designated CRO) will review the protocol and CRFs with the investigators and their staff. During the study, the field monitor will visit the site regularly to check the completeness of patient records, the accuracy of entries on the CRFs, the adherence to the protocol to Good Clinical Practice, the progress of enrollment, and to ensure that study treatment is being stored, dispensed, and accounted for according to specifications. Key study personnel must be available to assist the field monitor during these visits.

The investigator must maintain source documents for each patient in the study, consisting of case and visit notes (hospital or clinic medical records) containing demographic and medical information, laboratory data, electrocardiograms, and the results of any other tests or assessments. All information recorded on CRFs must be traceable to source documents in the patient's file. The investigator must also keep the original signed informed consent form (a signed copy is given to the patient).

The investigator must give the monitor access to all relevant source documents to confirm their consistency with the CRF entries. Novartis monitoring standards require full verification for the presence of informed consent, adherence to the inclusion/exclusion criteria and

documentation of SAEs. Additional checks of the consistency of the source data with the CRFs are performed according to the study-specific monitoring plan.

#### 9.3 Data collection

For studies using Electronic Data Capture (EDC), the designated investigator staff will enter the data required by the protocol into the Electronic Case Report Forms (eCRF). The eCRFs have been built using fully validated secure web-enabled software that conforms to 21 CFR Part 11 requirements, Investigator site staff will not be given access to the EDC system until they have been trained. Automatic validation programs check for data discrepancies in the eCRFs and, allow modification or verification of the entered data by the investigator staff.

The Principal Investigator is responsible for assuring that the data entered in eCRFs is complete, accurate, and that entry and updates are performed in a timely manner.

## 9.4 Database management and quality control

For studies using eCRFs, Novartis personnel (or designated CRO) will review the data entered by investigational staff for completeness and accuracy. Electronic data queries stating the nature of the problem and requesting clarification will be created for discrepancies and missing values and sent to the investigational site via the EDC system. Designated investigator site staff are required to respond promptly to queries and to make any necessary changes to the data.

At the conclusion of the study, the occurrence of any protocol violations will be determined. After these actions have been completed and the data has been verified to be complete and accurate, the database will be declared locked and made available for data analysis. Authorization is required prior to making any database changes to locked data, by joint written agreement between the Global Head of Biostatistics and Data Management and the Global Head of Clinical Development.

For EDC studies, after database lock, the investigator will receive a CD-ROM or paper copies of the patient data for archiving at the investigational site.

# 10 Statistical methods and data analysis

# 10.1 Analysis sets

The following sets will be used for statistical analysis and data reporting.

## 10.1.1 Full Analysis Set

Not applicable.

## 10.1.2 Safety set

The Safety Set includes all patients who received at least one dose of study medication after enrolling into the roll-over protocol.

#### 10.1.3 Dose-determining analysis set

Not applicable.

#### 10.2 Patient demographics/other baseline characteristics

Demographic and other baseline data characteristics will be summarized descriptively for the Safety Set.

## 10.3 Treatments (study treatment, compliance)

Dose administration data will be summarized using the Safety Set.

#### 10.4 Primary objective

The primary objective is to evaluate long term safety as assessed by the occurrence of AEs/SAEs.

#### 10.4.1 Variable

See Section 10.5.3.

#### 10.4.2 Statistical hypothesis, model, and method of analysis

No hypothesis will be tested.

## 10.4.3 Handling of missing values/censoring/discontinuations

Not applicable.

## 10.4.4 Supportive and Sensitivity analyses

No supportive analysis will be performed.

## 10.5 Secondary objectives

#### 10.5.1 Key secondary objective(s)

Not applicable.

## 10.5.2 Other secondary efficacy objectives

The secondary objective of the study is to evaluate clinical benefit as assessed by the investigator. Proportion of patients with clinical benefit as assessed by the investigator will be summarized at scheduled visits.

## 10.5.3 Safety objectives

The assessment of safety will be based mainly on the frequency of AEs and SAEs.

## 10.5.3.1 Analysis set and grouping for the analyses

The overall observation period will be divided into two mutually exclusive segments:

- 1. on-treatment period: from day of first dose of study medication in the roll-over study to 30 days after last dose of study medication
- 2. post-treatment period: starting at day 30+1 after last dose of study medication.

#### 10.5.3.2 Adverse events (AEs)

Summary tables for adverse events (AEs) will include only AEs that started or worsened during the on-treatment period, the *treatment-emergent* AEs. However, all safety data (including those from the post-treatment periods) will be listed and those collected during the post-treatment period are to be flagged.

The incidence of treatment-emergent adverse events (new or worsening from baseline) will be summarized by system organ class and or preferred term, severity (based on CTCAE grades), type of adverse event, relation to study treatment.

Deaths reportable as SAEs and non-fatal serious adverse events will be listed by patient and tabulated by type of adverse event.

#### 10.5.3.3 Other safety data

Not applicable.

#### 10.5.3.4 Supportive analyses for secondary

Not applicable.

#### 10.5.3.5 Tolerability

Not applicable.

#### 10.5.3.6 Pharmacokinetics

Not applicable.

## 10.6 Exploratory objectives

Not applicable.

#### 10.7 Interim analysis

Not applicable.

#### 10.8 Sample size calculation

Not applicable.

#### 10.9 Power for analysis of key secondary variables

Not applicable.

# 11 Ethical considerations and administrative procedures

#### 11.1 Regulatory and ethical compliance

This clinical study was designed, shall be implemented and reported in accordance with the ICH Harmonized Tripartite Guidelines for Good Clinical Practice, with applicable local regulations (including European Directive 2001/20/EC and US Code of Federal Regulations Title 21), and with the ethical principles laid down in the Declaration of Helsinki.

## 11.2 Responsibilities of the investigator and IRB/IEC/REB

The protocol and the proposed informed consent form must be reviewed and approved by a properly constituted Institutional Review Board/Independent Ethics Committee/Research Ethics Board (IRB/IEC/REB) before study start. Prior to study start, the investigator is required to sign a protocol signature page confirming his/her agreement to conduct the study in accordance with these documents and all of the instructions and procedures found in this protocol and to give access to all relevant data and records to Novartis monitors, auditors, Novartis Clinical Quality Assurance representatives, designated agents of Novartis, IRBs/IECs/REBs and regulatory authorities as required.

## 11.3 Informed consent procedures

Eligible patients may only be included in the study after providing written (witnessed, where required by law or regulation), IRB/IEC/REB-approved informed consent

Informed consent must be obtained before conducting any study-specific procedures (i.e. all of the procedures described in the protocol). The process of obtaining informed consent should be documented in the patient source documents. The date when a subject's Informed Consent was actually obtained will be captured in their CRFs.

Novartis will provide to investigators, in a separate document, a proposed informed consent form (ICF) that is considered appropriate for this study and complies with the ICH GCP guideline and regulatory requirements. Any changes to this ICF suggested by the investigator must be agreed to by Novartis before submission to the IRB/IEC/REB, and a copy of the approved version must be provided to the Novartis monitor after IRB/IEC/REB approval.

Women of child bearing potential should be informed that taking the study medication may involve unknown risks to the fetus if pregnancy were to occur during the study and agree that in order to participate in the study they must adhere to the contraception requirement for the duration of the study. If there is any question that the patient will not reliably comply, they should not be entered in the study.

#### Additional consent form

Not applicable.

# 11.4 Discontinuation of the study

Novartis reserves the right to discontinue this study under the conditions specified in the clinical study agreement. Specific conditions for terminating the study are outlined in Section 4.4.

#### 11.5 Publication of study protocol and results

Novartis assures that the key design elements of this protocol will be posted in a publicly accessible database such as clinicaltrials.gov. In addition, upon study completion and finalization of the study report the results of this study will be either submitted for publication and/or posted in a publicly accessible database of clinical study results.

# 11.6 Study documentation, record keeping and retention of documents

Each participating site will maintain appropriate medical and research records for this trial, in compliance with Section 4.9 of the ICH E6 GCP, and regulatory and institutional requirements for the protection of confidentiality of subjects. As part of participating in a Novartis-sponsored study, each site will permit authorized representatives of the sponsor(s) and regulatory agencies to examine (and when required by applicable law, to copy) clinical records for the purposes of quality assurance reviews, audits and evaluation of the study safety and progress.

Source data are all information, original records of clinical findings, observations, or other activities in a clinical trial necessary for the reconstruction and evaluation of the trial. Examples of these original documents and data records include, but are not limited to, hospital records, clinical and office charts, laboratory notes, memoranda, subjects' diaries or evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies or transcriptions certified after verification as being accurate and complete, microfiches, photographic negatives, microfilm or magnetic media, x-rays, and subject files and records kept at the pharmacy, at the laboratories, and medico-technical departments involved in the clinical trial.

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site Principal Investigator. The study case report form (CRF) is the primary data collection instrument for the study. The investigator should ensure the accuracy, completeness, legibility, and timeliness of the data reported in the CRFs and all other required reports. Data reported on the CRF, that are derived from source documents, should be consistent with the source documents or the discrepancies should be explained. All data requested on the CRF must be recorded. Any missing data must be explained. Any change or correction to a paper CRF should be dated, initialed, and explained (if necessary) and should not obscure the original entry. For electronic CRFs an audit trail will be maintained by the system. The investigator should retain records of the changes and corrections to paper CRFs.

The investigator/institution should maintain the trial documents as specified in Essential Documents for the Conduct of a Clinical Trial (ICH E6 Section 8) and as required by applicable regulations and/or guidelines. The investigator/institution should take measures to prevent accidental or premature destruction of these documents.

Essential documents (written and electronic) should be retained for a period of not less than fifteen (15) years from the completion of the Clinical Trial unless Sponsor provides written permission to dispose of them or, requires their retention for an additional period of time because of applicable laws, regulations and/or guidelines.

#### 11.7 Confidentiality of study documents and patient records

The investigator must ensure anonymity of the patients; patients must not be identified by names in any documents submitted to Novartis. Signed informed consent forms and patient enrollment log must be kept strictly confidential to enable patient identification at the site.

## 11.8 Audits and inspections

Source data/documents must be available to inspections by Novartis or designee or Health Authorities.

#### 11.9 Financial disclosures

Financial disclosures should be provided by study personnel who are directly involved in the treatment or evaluation of patients at the site - prior to study start.

#### 12 Protocol adherence

Investigators ascertain they will apply due diligence to avoid protocol deviations. Under no circumstances should the investigator contact Novartis or its agents, if any, monitoring the study to request approval of a protocol deviation, as no authorized deviations are permitted. If the investigator feels a protocol deviation would improve the conduct of the study this must be considered a protocol amendment, and unless such an amendment is agreed upon by Novartis and approved by the IRB/IEC/REB it cannot be implemented. All significant protocol deviations will be recorded and reported in the CSR.

# 12.1 Amendments to the protocol

Any change or addition to the protocol can only be made in a written protocol amendment that must be approved by Novartis, Health Authorities where required, and the IRB/IEC/REB. Only amendments that are required for patient safety may be implemented prior to IRB/IEC/REB approval. Notwithstanding the need for approval of formal protocol amendments, the investigator is expected to take any immediate action required for the safety of any patient included in this study, even if this action represents a deviation from the protocol. In such cases, Novartis should be notified of this action and the IRB/IEC at the study site should be informed according to local regulations (e.g. UK requires the notification of urgent safety measures within 3 days) but not later than 10 working days.

# 13 References (available upon request)

Boulay A, Lane HA (2007) The mammalian target of rapamycin kinase and tumor growth inhibition. Recent Results Cancer Res. 2007;172:99-124.

Krishna G, Moton A, Lei Ma L, et al (2009) Effects of oral posaconazole on the pharmacokinetic properties of oral and intravenous midazolam: A phase I, randomized, openlabel, crossover study in healthy volunteers. Clinical Therapeutics; 31(2): 286-98.